CLINICAL TRIAL: NCT03277014
Title: Insulin-like Growth Factor-1 as a Nutritional Monitoring Factor in Patients With Chronic Intestinal Failure
Brief Title: Using IGF-1 for Nutritional Monitoring
Status: Completed | Type: Observational
Sponsor: Wang Xinying (Other)
Responsible Party: Sponsor-Investigator, Wang Xinying, Director of the clinical nutrition center, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Other Study IDs: 201502022-3
Record Dates: First submitted 2017-09-03; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Nutritional Supplement
Keywords: Nutritional monitoring; insulin-like growth factor-1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nutrition support is critical to a vast number of patients who are hospitalized annually because of critical illnesses or surgery. It is also necessary for patients with chronic intestinal failure (CIF), who often require parenteral nutrition over periods of weeks or months. While scoring systems that assess nutritional risks in patients exist, there are no guidelines for continuous nutritional monitoring during supplementation and parenteral feeding. Previous studies have hinted that insulin-like growth factor-1 (IGF-1) may serve as a biomarker for nutritional support efficiency; however, such studies were not statistically definitive. Therefore, the investigators aimed to assess IGF-1 as a biomarker for both diagnosing nutritional risk and malnutrition and for monitoring the efficiency of nutritional support, particularly compared to other biomarkers such as BMI as well as albumin, prealbumin, transferrin, and retinol-binding protein.

DETAILED DESCRIPTION:
Chronic intestinal failure (CIF) is one of the rarest of organ failures all over the world, mainly caused by severe gastrointestinal or systemic benign diseases such as intestinal ﬁstula, short bowel, and mechanical obstruction. Moreover, patients with end-stage intra-abdominal or pelvic cancer can also develop into CIF. CIF is deﬁned as gut function that is below the minimum necessary for the absorption of macronutrients and/or water and electrolytes; in such cases, nutrition support, especially for parenteral nutrition, is indispensable to maintain health and recovery for CIF patients.

Nutrition support has successfully saved the lives of thousands of patients with CIF, as well as those who have critical illnesses or underwent surgery. According to the guidelines, patients with CIF require parenteral nutrition over periods of weeks or months and the efficiency of nutrition support will influence the prognoses directly . The exact nutritional assessment and close nutritional monitoring are key points to optimize nutritional therapy. Firstly, the recommended scoring systems such as the Nutritional Risk Screening 2002 (NRS-2002) score or the 'nutrition risk in the critically ill' (NUTRIC) score can identify patients who are at nutritional risk and who would benefit from nutritional support. Secondly, nutritional support regimens should be individualized and adjusted over time based on continuous monitoring; however, there are no guidelines regarding such nutritional monitoring. The NRS-2002 and NUTRIC scores are recommended as initial nutritional assessment indices, but are inappropriate for continuous evaluation. Moreover, validated biomarkers that can be used for monitoring short-term nutritional status changes were still unclear. Nowadays, common serum protein markers such like albumin, prealbumin, transferrin, and retinol-binding protein (RBP) are used to monitor the efficiency of nutritional support in clinical practice [5, 8]. However, all these biomarkers failed to reflect changes of nutritional status with sufficient sensitivity in CIF patients.

Insulin-like growth factor-1 (IGF-1) is an IGF family member that consists of 70 amino acid residues. IGF-I was first reported as a nutritional marker in 1973 because its serum concentrations are reduced during malnutrition; its serum levels also proved to be affected by protein or/and energy deficiency. Several previous studies reported that IGF-1 is a more sensitive and speciﬁc indicator of nutritional status than prealbumin, transferrin, or RBP because of its shorter serum half-life and more accurate response to nutritional intake; however, these studies had small cohorts.

In present study, the investigators compared IGF-1 to traditional serum biomarkers in terms of diagnosing nutritional risk and malnutrition, as well as in monitoring the efficiency of nutrition support in CIF patients.

the investigators conducted a retrospective study of patients treated at a single clinical nutrition center of a tertiary referral hospital in China to investigate whether the measurement of IGF-1 is useful for monitoring the efficiency of nutritional support and to explore the relationship between IGF-1 and lean body mass in CIF patients. The influence of IGF-1 was also explored in this study. The data used were accumulated at the center between September 2013 and January 2017. All adult CIF patients (age ≥18 years) receiving nutrition support were included. The exclusion criteria were hepatic insufficiency (alanine transaminase/aspartate transaminase ratio 200% above normal range or bilirubin >3 mg/dL), renal insufficiency (serum creatinine [Scr] >1.5 mg/dL), acute or life-threatening diseases (e.g., shock, collapse, stroke, coma of unknown etiology, or recent cardiac infarction), and pregnant or breast-feeding women. The study was approved by the ethics committee of Jinling Hospital, Medical School of Nanjing University.

Malnutrition was defined as weight loss >10% within 6 months, a body mass index (BMI) <18.5, a subjective global assessment (SGA) score of stage C, or albumin level <30 g/L. Serum IGF-1, albumin, pre-albumin, transferrin, RBP, creatinine, and hemoglobin were measured weekly in patients receiving nutrition support after hospital admission. The resting energy expenditure, predicted weekly by indirect calorimetry (Quark PFT ERGO , COSMED Srl - Italy), was used to guide energy delivery. The target dose of protein intake was 1.2 g/kg/day, which was adjusted according to the level of serum albumin. Patients were also subjected to strict fluid intake management. The nutritional support schemes were recorded daily, and the body composition was also measured weekly to estimate nutrition status (Inbody S10, Biospace).

ELIGIBILITY:
Inclusion Criteria:

* All adult CIF patients (age ≥18 years) receiving nutrition support were included

Exclusion Criteria:

* Hepatic insufficiency (alanine transaminase/aspartate transaminase ratio 200% above normal range or bilirubin >3 mg/dL), renal insufficiency (serum creatinine [Scr] >1.5 mg/dL), acute or life-threatening diseases (e.g., shock, collapse, stroke, coma of unknown etiology, or recent cardiac infarction), and pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at a single clinical nutrition center of a tertiary referral hospital in China to investigate whether the measurement of IGF-1 is useful for monitoring the efficiency of nutritional support and to explore the relationship between IGF-1 and lean body mass in CIF patients. The data used were accumulated at the center between September 2013 and January 2017.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Nutrition indicators | From date of patients enrollment until the date of patients discharge from hospital, assessed up to 2 months.
  Insulin-like growth factor-1/Hemoglobin/albumin/prealbumin/transferrin/retinol binding protein/serum creatinine/cholesterol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Bielawska B, Allard JP. Nutrients 2017, 9(5). 2. Pironi L, Arends J, Bozzetti F, Cuerda C, Gillanders L, Jeppesen PB, Joly F, Kelly D, Lal S, Staun M et al. Clinical nutrition 2016, 35(2):247-307. 3. Pironi L. Best Pract Res Clin Gastroenterol 2016, 30(2):173-185. 4. Feinberg J, Nielsen EE, Korang SK, Halberg Engell K, Nielsen MS, Zhang K, Didriksen M, Lund L, Lindahl N, Hallum S et al. The Cochrane database of systematic reviews 2017, 5:Cd011598. 5. Taylor BE, McClave SA, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA et al. Crit Care Med 2016, 44(2):390-438. 6. McClave SA, DiBaise JK, Mullin GE, Martindale RG. Am J Gastroenterol 2016, 111(3):315-334.
- [Derived] Wang P, Yang J, Zhang Y, Zhang L, Gao X, Wang X. Risk Factors for Renal Impairment in Adult Patients With Short Bowel Syndrome. Front Nutr. 2021 Jan 18;7:618758. doi: 10.3389/fnut.2020.618758. eCollection 2020. PMID 33537339
- [Derived] Wang X, Tian F, Sun H, Zhang L, Gao X, Huang Y, Yang J, Shen R, Wang J, Jiang T, Chen P, Liu S, Li J. Insulin-like growth factor-1 as a nutritional monitoring factor in patients with chronic intestinal failure. Clin Nutr. 2019 Aug;38(4):1737-1744. doi: 10.1016/j.clnu.2018.07.031. Epub 2018 Aug 2. PMID 30126709